CLINICAL TRIAL: NCT05512429
Title: Prognostic Value of Body Composition in Therapy-Naïve Patients With Non-Small Cell Lung Cancer
Brief Title: Prognostic Value of Body Composition in Lung Cancer
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2019.1026
Record Dates: First submitted 2022-08-18; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Body Composition and Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stage-IV non small cell lung cancer (NSCLC): Eighty-three patients with stage-IV NSCLC who received at least one cycle of platinum based chemotherapy (PBCT) or tyrosine kinase inhibitor (TKI) therapy and who underwent pre treatment fluorodeoxyglucose (FDG)-positron emission tomography (PET) /computed tomography (FDG PET/CT) from June 2012 to February 2019
  Interventions: Other: measured of body composition with computed tomography

INTERVENTIONS:
Other: measured of body composition with computed tomography — Multislice and single-slice computed tomography images were used for assessment of body composition including visceral adipose tissue (VAT), subcutaneous adipose tissue (SAT), skeletal muscle mass volume (SMMV)

SUMMARY:
The effect of body composition on the survival rate is one of the research topics of interest in cancer patients and gaining attention in the last years. Body mass index is often used a proxy measure of total adiposity and previous studies examining the relationship between BMI and cancer outcomes have been showed distinct results . Obese patients with malignancies such as colorectal, breast, and pancreatic cancers, have been shown to have a worse prognosis than normal-weight patients . Nevertheless, obese patients with non small cell lung cancer(NSCLC) have been observed to have a better clinical outcome than normal/low-weight cancer patients . In this study, we examined the effects of subcutaneous adipose tissue, visceral adipose tissue and skeletal muscle volumes on survival in metastatic NSCLC patients under different treatment regimens. Since there is no standard method for adipose tissue measurement, we evaluated the abdominal cavity with multi-slice and single-slice computed tomography measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Having a pathological diagnosis of non small cell lung cancer
2. Having a stage-IV disease
3. To have received at least one course of treatment
4. Presence of positron emission tomography /computed tomography (PET/CT) examination before treatment and having it taken in our hospital
5. The data about the study can be accessed in our center.
6. To be over 18 years old

Exclusion Criteria:

1. Unable to access patients data
2. PET/CT CDs cannot be accessed or are not suitable for evaluation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eighty-three patients with stage-IV NSCLC who received at least one cycle of platinum based chemotherapy (PBCT) or tyrosine kinase inhibitor (TKI) therapy and who underwent pre treatment FDG PET/CT from June 2012 to February 2019
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the impact of visceral adipose tissue (VAT) on the prognosis of metastatic non-small cell lung cancer (NSCLC) patients. | through study completion, an average of 6 months
  Visceral adipose tissue (VAT) area was measured by using computed tomography (CT). The entire abdominopelvic region from the "diaphragm dome" to the "symphysis pubis" level was determined as the study area. The volume was recorded as cm3. Index values were calculated by proportioning VAT to body surface area (BSA) and median index value was determined. The survival rates of patients with an index value greater and less than the mean index value were compared.
To evaluate the impact of subcutaneous adipose tissue (SAT) on the prognosis of metastatic non-small cell lung cancer (NSCLC) patients. | through study completion, an average of 6 months
  Subcutaneous adipose tissue (SAT) area was measured by using computed tomography (CT). The entire abdominopelvic region from the "diaphragm dome" to the "symphysis pubis" level was determined as the study area. The volume was recorded as cm3. Index values were calculated by proportioning SAT to body surface area (BSA) and median index value was determined. The survival rates of patients with an index value greater and less than the mean index value were compared.
To evaluate the impact of skeletal muscle mass volume (SMMV) on the prognosis of metastatic non-small cell lung cancer (NSCLC) patients. | through study completion, an average of 6 months
  Skeletal muscle mass volume (SMMV) area was measured by using computed tomography (CT). For SMMV calculation, paraspinal muscle tissue located between L2-L5 lumbar vertebrae levels was determined . The volume was recorded as cm3. Index values were calculated by proportioning SMMV to body surface area (BSA) and median index value was determined. The survival rates of patients with an index value greater and less than the mean index value were compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Tuğba Kıratlı Yolcu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No